CLINICAL TRIAL: NCT05093270
Title: A First-in-Human, Single- and Multiple-Ascending Dose and Food-Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BGB-23339 in Healthy Subjects
Brief Title: First-in-Human, Single- and Multiple-Ascending Dose and Food-Effect Study of BGB-23339 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BGB-23339-101
Record Dates: First submitted 2021-09-16; First posted 2021-10-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Not Determined

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A Dose Escalation (Single Ascending Dose) (Experimental): Up to 5 dose levels of BGB-23339 or Placebo
  Interventions: Drug: BGB-23339; Drug: Placebo
- Part B Dose Escalation (Multiple Ascending Dose) (Experimental): Up to 4 dose levels of BGB-23339 or placebo based on data collected in Part A
  Interventions: Drug: BGB-23339; Drug: Placebo
- Part C Dose Escalation (Multiple Ascending Dose in Chinese Subjects Sub-study) (Experimental): Up to 2 dose levels of BGB-23339 or placebo based on data collected in Part A and B (conducted in China only)
  Interventions: Drug: BGB-23339; Drug: Placebo
- Part D (Food-Effect Study) (Experimental): Three single dose levels of BGB-23339 under different feeding conditions
  Interventions: Drug: BGB-23339

INTERVENTIONS:
Drug: BGB-23339 — Administered orally as a tablet
Drug: Placebo — Administered orally as a tablet
  Arms: Part A Dose Escalation (Single Ascending Dose); Part B Dose Escalation (Multiple Ascending Dose); Part C Dose Escalation (Multiple Ascending Dose in Chinese Subjects Sub-study)

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of BGB-23339 and food effects in healthy participants

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) and able to comply with study requirements
2. Healthy men and/or women of no childbearing potential of age ≥ 18 years and ≤ 55 years on the day of signing the ICF (or the legal age of consent) for Parts A, B and D; of age≥ 18 years and ≤ 45 years on the day of signing the ICF (or the legal age of consent) and of Chinese descent for Part C
3. Participants are in good general health as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring
4. Body weight ≥ 50 kg and body mass index (BMI) within the range 18 to 32 kg/m2 (inclusive)
5. A nonsterile man with a female partner of childbearing potential must be willing to use a highly effective method of birth control from the time of study enrollment until 90 days after the last dose of study drug
6. A woman of no childbearing potential must meet at least one of the following criteria:

   1. Postmenopausal status, defined as: cessation of regular menses for ≥ 12 consecutive months (menopause confirmed by Follicular Stimulating Hormone [FSH] levels and Luteinizing Hormone [LH] levels as defined by the established reference ranges)
   2. Surgically sterile (eg, hysterectomy, oophorectomy, or tubal ligation for at least the past 3 months).

Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug; or interfering with the interpretation of data
2. Abnormal blood pressure as determined by the investigator
3. Active herpes infection, including herpes simplex 1 and 2 and herpes zoster (demonstrated on physical examination and/or medical history ≤ 2 months before randomization)
4. Any malignancies within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
5. Past or intended use of prescription medication ≤ 14 days and over-the-counter (OTC) medication including herbal, vitamins and dietary supplements ≤ 7 days before randomization
6. Live vaccine ≤ 30 days, and/or vaccine of any type ≤ 14 days before randomization
7. Has received an investigational product within the following time before randomization: 3 months, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer)
8. Participation in a prior study that would result in loss of blood or blood products in excess of 500 mL within 56 days before randomization
9. Exposure to ≥ 4 new chemical entities within 12 months before randomization
10. Presence of hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) at screening or ≤ 3 months before randomization
11. Regular alcohol consumption ≤ 3 months before randomization
12. Regular use of recreational drugs
13. Current use and/or has used nicotine or nicotine-containing products (eg, nicotine patch and electronic cigarette) within 14 days before randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 7 weeks
Number of participants with clinically significant changes from baseline in vital signs | Up to approximately 4 weeks
  Vital signs include blood pressure and pulse rate
Number of participants with clinically significant changes from baseline in clinical laboratory values | Up to approximately 4 weeks
  Laboratory values include hematology, clinical chemistry, coagulation, and urinalysis

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to last quantifiable time (AUClast) for Parts A, B, C and D | Up to approximately 4 weeks
Area under the plasma concentration-time curve from time zero to 24 hours postdose (AUC0-24) for Part D only | Up to approximately 4 weeks
Area under the plasma concentration-time curve from time zero to end of dosing interval (AUCtau) for Parts A, B, C and D | Up to approximately 4 weeks
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) for Parts A, B, C, and D | Up to approximately 4 weeks
Maximum observed plasma concentration (Cmax) for Parts A, B, C and D | Up to approximately 4 weeks
Time to maximum plasma concentration (Tmax) for Parts A, B, C and D | Up to approximately 4 weeks
Trough plasma concentration (Ctrough) for Parts A, B, and C | Up to approximately 4 weeks
Apparent terminal elimination half-life (t½) for Parts A, B, C and D | Up to approximately 4 weeks
  in fed and fasted states for BGB-23339
Apparent systemic clearance (CL/F) for Parts A, B, and C | Up to approximately 4 weeks
Apparent volume of distribution (Vz/F) for Parts A, B, and C | Up to approximately 4 weeks
Accumulation ratios, and metabolite to parent ratio for BGB-23339 and its metabolite BGB-25808 as appropriate for Parts A, B, C and D | Up to approximately 4 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Q PHARM, Herston, Queensland
  - Nucleus Network, Melbourne, Victoria
- The Affiliated Hospital of Qingdao University Branch West Coast, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes